CLINICAL TRIAL: NCT04853537
Title: Impact of Intermittent Fasting on the Incidence of Gestational Diabetes Mellitus(DM) in Obese Pregnant Women in 3rd Trimester
Brief Title: Intermittent Fasting on the Incidence of Gestational Diabetes Mellitus Obese Pregnant Women in 3rd Trimester
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: effect of IF on GD in obese
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-04

CONDITIONS: Intermittent Fasting; Gestational Diabetes; Obesity
MeSH Terms: conditions — Intermittent Fasting; Diabetes, Gestational; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): • 126 women will fast 16 consecutive hours per day including sleeping hours. and follow them from 26w till 36w by GTT(glucose tolerance test) and the weight gain and incidence of gestational diabetes
  Interventions: Dietary Supplement: intermittent fasting diet
- control group (No Intervention): • 126 women will not fasting with the same life style and follow the incidence of gestational diabetes

INTERVENTIONS:
Dietary Supplement: intermittent fasting diet — intermittent fasting diet to obese pregnant women >30 BMI and incidence of gestational diabetes
  Arms: study group

SUMMARY:
This randomized controlled clinical trial will assess the impact of intermittent fasting on the incidence of gestational DM in obese pregnant women in 3rd trimester and its effect on maternal and neonatal outcomes.

DETAILED DESCRIPTION:
The term intermittent fasting, when used for health reasons or weight loss, has been used to describe various types of caloric restriction. Some authors use it when a patient withholds caloric intake for several consecutive hours during the day (often 16 h with all energy intake during the other 8 h of the day, others for a full day once or twice a week , and others three or four days per week Some protocols allow protein intake but no carbohydrates and still label it intermittent fasting.

Others allow carbohydrates or macro/micro-nutrients up to a limit that will still promote ketosis and, although it is simply a low-calorie diet, due to the popularity of fasting this has been labeled a diet that mimics fasting.

In this protocol we use 16hour fasting in 24hour with the same caloric intake in 8hour and can drink water ,coffee , and other noncaloric beverages during the fast, which can help reduce feelings of hunger .

In all instances, non-caloric fluid intake is permitted (which is one of the main differences when compared to religious fasting) and therefore significantly reduces the risk of dehydration and hypotension, a prominent consideration in religious fasting.

During the fasting hours and after breaking the fast, metabolic condition of the body could be influenced as a consequence of change in the pattern and amount of activity, meals and fluid intake, and even sleeping hours.

Intermittent fasting and low caloric intake have been shown to improve various metabolic and inflammatory pathways. Insulin resistance, the most prominent feature of type 2 diabetes during pregnancy, has long been known to improve with intermittent fasting. After a period of fasting, insulin sensitivity rises and insulin levels fall. These result in improved fasting and postprandial glucose levels. In addition, as insulin induces adipose tissue growth, there is less propensity to weight gain and potentially even weight loss which leading to decrease neonatal adverse effects of gestational DM and improved fetal outcome.

On the other hand, many other studies found that fasting has no effect on intrauterine growth, birth weight, birth-time indices, gestational diabetes, preterm birth, and preeclampsia. Predominantly, results of the studies examining the effects of fasting on mothers and newborns are not homogenous; therefore, further research should be conducted to attain valid findings.

ELIGIBILITY:
Inclusion Criteria:

- 1. Healthy pregnant women. 2. Age (18 - 35 years old). 3. Women with BMI (_> 30 kg/m2).

4. A living singleton pregnancy. Gestational age (24- 27 weeks).(recruitment time)

Exclusion Criteria:

- 1. Multiple gestations. 2. Women with diabetes 3. pre-pregnancy cardiovascular disease, chronic hypertensive, and pregnancy-induced hypertension; blood pressure _> 140/90.

4. Women with hepatic, renal diseases or coagulopathy 5. Women with peptic ulcer.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
gestational diabetes | from 24-36 weeks of gestation
  percentage of diabetes in obese patient is increased by 1.3% and it will be assessed by glucose tolerance test

SECONDARY OUTCOMES:
Maternal weight gain, | from 24-36 weeks of gestation
  maternal
Fetal weight | on labour
  fetal out come during delivery
fetal Apgar score | on labour
  score for baby after labour
NICU(neonatal intensive care unit) admission | on labour
  fetal
mode of delivery | on 36 weeks of gestation
  NVD NVD(normal vaginal delivery) or C.S(caesarian section)
any associated comorbidities questionnaires | from 24-36 weeks of gestation
  if there is other diseases developed like gestational hypertension

CONTACTS AND LOCATIONS:
Overall Officials: reda mokhtar, lecuterer, Principal Investigator — Ain Shams University

REFERENCES:
- [Background] Alkandari JR, Maughan RJ, Roky R, Aziz AR, Karli U. The implications of Ramadan fasting for human health and well-being. J Sports Sci. 2012;30 Suppl 1:S9-19. doi: 10.1080/02640414.2012.698298. Epub 2012 Jun 29. PMID 22742901
- [Background] Carter S, Clifton PM, Keogh JB. Effect of Intermittent Compared With Continuous Energy Restricted Diet on Glycemic Control in Patients With Type 2 Diabetes: A Randomized Noninferiority Trial. JAMA Netw Open. 2018 Jul 6;1(3):e180756. doi: 10.1001/jamanetworkopen.2018.0756. PMID 30646030
- [Background] Corley BT, Carroll RW, Hall RM, Weatherall M, Parry-Strong A, Krebs JD. Intermittent fasting in Type 2 diabetes mellitus and the risk of hypoglycaemia: a randomized controlled trial. Diabet Med. 2018 May;35(5):588-594. doi: 10.1111/dme.13595. Epub 2018 Feb 27. PMID 29405359
- [Background] Furmli S, Elmasry R, Ramos M, Fung J. Therapeutic use of intermittent fasting for people with type 2 diabetes as an alternative to insulin. BMJ Case Rep. 2018 Oct 9;2018:bcr2017221854. doi: 10.1136/bcr-2017-221854. PMID 30301822
- [Background] Grajower MM, Horne BD. Clinical Management of Intermittent Fasting in Patients with Diabetes Mellitus. Nutrients. 2019 Apr 18;11(4):873. doi: 10.3390/nu11040873. PMID 31003482
- [Background] Kim SY, England L, Wilson HG, Bish C, Satten GA, Dietz P. Percentage of gestational diabetes mellitus attributable to overweight and obesity. Am J Public Health. 2010 Jun;100(6):1047-52. doi: 10.2105/AJPH.2009.172890. Epub 2010 Apr 15. PMID 20395581
- [Background] Harris L, Hamilton S, Azevedo LB, Olajide J, De Brun C, Waller G, Whittaker V, Sharp T, Lean M, Hankey C, Ells L. Intermittent fasting interventions for treatment of overweight and obesity in adults: a systematic review and meta-analysis. JBI Database System Rev Implement Rep. 2018 Feb;16(2):507-547. doi: 10.11124/JBISRIR-2016-003248. PMID 29419624
- [Background] Klempel MC, Kroeger CM, Bhutani S, Trepanowski JF, Varady KA. Intermittent fasting combined with calorie restriction is effective for weight loss and cardio-protection in obese women. Nutr J. 2012 Nov 21;11:98. doi: 10.1186/1475-2891-11-98. PMID 23171320
- [Background] Sakar MN, Gultekin H, Demir B, Bakir VL, Balsak D, Vuruskan E, Acar H, Yucel O, Yayla M. Ramadan fasting and pregnancy: implications for fetal development in summer season. J Perinat Med. 2015 May;43(3):319-23. doi: 10.1515/jpm-2013-0289. PMID 24810552
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779